CLINICAL TRIAL: NCT00930241
Title: Prospective Randomized Trial to Compare a Twice Daily to a Once Daily Administration of the Tacrolimus in Lung Transplanted Patients
Brief Title: Twice Daily Versus Once Daily Administration of the Tacrolimus in Lung Transplantation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: logistic reasons (insufficient funding, technical problems with MEMS)
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5281M mono
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Lung Transplantation
Keywords: Lung Transplantation; Tacrolimus; Deterioration of graft function
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advagraf (Experimental): Advagraf® (one daily dose of Tacrolimus)
  Interventions: Drug: Advagraf®
- Prograf (Active Comparator): Prograf® (two daily doses of Tacrolimus)
  Interventions: Drug: Prograf®

INTERVENTIONS:
Drug: Advagraf® — Advagraf® (one daily dose of Tacrolimus)
  Arms: Advagraf
Drug: Prograf® — Prograf® (two daily doses of Tacrolimus)
  Arms: Prograf

SUMMARY:
This study is a prospective randomized trial to compare twice daily to once daily administration of the basic immunosuppressive regimen in lung transplanted patients.

DETAILED DESCRIPTION:
Prevalence data of non-compliance in solid organ transplantations fluctuate is reported in up to 39% of transplant recipients (z. B. for lung transplantations 13 - 22%; Kugler et al.). Non-compliance with immunosuppressive therapy is associated with an increased risk of late-acute rejections and the development of chronic transplant dysfunction. Chronic transplant dysfunction (bronchiolitis obliterans- syndrome-BOS) is the second most causing for organ failure after the first year following lung transplantation and often leads to re-transplantation or death. Preventative procedures for improving the compliance are simplification of the dose of the immunosuppressants (a once daily dose instead of a twice daily dose), the prescription of an immunosuppressants with less side-effects and to raise the patient´s awareness for having the greatest responsibility for the efficacy of his therapy. Prospective studies and metaanalysis revealed that the probability for a good compliance can be more than doubled at once daily administration in comparison to twice daily and the best predictor for a good compliance is an easy therapy. For this reason we want to investigate the extent of profit for our lung transplant patients receiving once daily basis immunosuppression in comparison to those who receive twice daily dose.

Hypothesis: Patients of the once daily administration group of the immunosuppressive medication will have a better compliance compared to the twice daily group (as measured by the endpoints variability and medication abstraction from the electronic devices)

ELIGIBILITY:
Inclusion Criteria:

* Patients (Pts) more than 1 year after single lung, double lung or heart/lung transplantation
* Pts treated with cyclosporin, steroids and MMF
* Pts ≥ 18 and ≤ 70 years and
* Pts with one of the following:

  * pts with recurrent acute rejections (RAR)
  * two or more acute rejections in 3 months (first 3 years post Tx, 6 months (> 3 years post Tx) defined by:

    * transbronchial biopsy > A1 (or A1 with clinical criteria below) nach ISHLT (B>1R) or
    * decline of FEV1 > 10 % baseline after exclusion of infection, airway complication, effusion etc. and improvement to steroid-pulse therapy (methylprednisolone 15 mg/kg for three days) = FEV1 improvement > 10% compared to the last measurement before AR treatment
* Pts with steroid-resistant or ongoing acute rejections (OAR) defined by:

  * transbronchial biopsy > A1 (or A1 with clinical criteria above) at least 4 weeks following steroid-pulse therapy (methylprednisolone 15 mg/kg for three days) or
  * no FEV1 improvement (< 5% baseline) at least 14 days following ACR steroid-pulse therapy (methylprednisolone 15 mg/kg for three days) after exclusion of infection, airway complication, effusion etc. or
* Pts with new onset of BOS (nBOS) Unexplained FEV1 < 80% of baseline after exclusion of Infection, airway complication, effusion etc
* Pts with CyA associated side effects (e.g., hyperlipidaemia, hypertriglyceridemia, hypertension, hirsutism, gingival hyperplasia)

Exclusion Criteria:

* Pregnant or breast feeding women
* Pts who are not using a double-barrier method of birth control
* Pts with systemic infections
* Pts with severe diarrhea, vomiting, active ulcer
* Pts with severe liver disease or liver cirrhosis
* Pts with m-Tor inhibitors
* Pts with hypersensitivity to Tacrolimus, other macrolides or other tablet ingredients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Improvement of adherence as measured by Tacrolimus trough level below the target level and dispensing of less than 50% of the prescribed doses in the last three days measured electronically before this subtherapeutic drug monitoring | 6 months

SECONDARY OUTCOMES:
Deterioration of graft function (FEV1) before and at month 12 after conversion | 6 months
Number of drug holidays (intake of less than 50% of prescribed doses in 24 hours) measured electronically | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens T Gottlieb, M.D., Principal Investigator — Hannover Medical School
Locations (3):
- Germany (3):
  - Department of Respiratory Medicine, Medizinische Hochschule Hannover, Hanover
  - Hannover Medical School, Dept. of Respiratory Medicine, Hanover
  - Hannover Medical School, Hanover